CLINICAL TRIAL: NCT01380236
Title: A Phase II, Two-centre, Single Blind Study to Evaluate the Safety, Tolerability and Explore the Efficacy of 8.0 mg ASM8 Inhaled Daily for 14 Days in Adult Subjects With Moderate to Severe Asthma
Brief Title: A Single Blind Study to Evaluate the Safety, Tolerability and Explore the Efficacy of 8.0 mg ASM8 Inhaled Daily for 14 Days in Severe Asthma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol not progressed. Study not implemented.
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ASM8-A-208
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ASM8

SUMMARY:
The purpose of the study is to determine the safety and tolerability of 8.0 mg of ASM8 when given daily for 14 days by the Aeroneb® Go nebulizer to subjects with moderate to severe asthma.

DETAILED DESCRIPTION:
The safety and tolerability of ASM8 will be assessed by performing a physical exam and vital signs, measuring the use of concomitant medication, routine laboratory tests, urinalysis, sputum analysis, serum IL-1 and TNF-α, lung carbon monoxide diffusion capacity, pulse oximetry and measuring AEs

There are 5 study phases: screening (phase 1), run-in (phase 2), treatment A (phase 3) with Active or Placebo, treatment B(phase 4) with Active or Placebo and end of study (phase 5) that includes a wash out period and a final visit.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with asthma for 3 or more months Have moderate to severe asthma as defined by ATS criteria

Exclusion Criteria:

* No history of pulmonary or health problems for which the Investigator considers that participation in this protocol is a risk for the subject

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Sputum total cells, differential and sputum levels of IL-1 and TNF alpha | 56 days
  Sputum total cells, differential (neutrophils, macrophages, bronchial cells and lymphocytes) and sputum levels of IL-1 and TNF alpha at the end of each treatment and at the final visit will be reported as absolute counts (10x6 cells/mL) and percentages (%) and change in % from baseline will also be presented.